CLINICAL TRIAL: NCT05603416
Title: Investigation of Benegut® on Immediate GI Discomfort Relief Caused by Acute Overfeeding in Healthy Subjects- a Randomized, Placebo-controlled Cross-over Study
Brief Title: Investigation of Benegut® on Immediate GI Discomfort Relief Caused by Acute Overfeeding in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vital Solutions GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: BTS1308/19
Record Dates: First submitted 2022-10-21; First posted 2022-11-02 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Digestive health; Perilla frutescens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benegut (Active Comparator): Dietary Supplement: Perilla frutescens extract
  Interventions: Dietary Supplement: Perilla frutescens extract
- Placebo (Placebo Comparator): Dietary Supplement: Placebo, no active ingredient
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Perilla frutescens extract — oral dissolvable powder - dosage 300mg
  Arms: Benegut
Dietary Supplement: Placebo — oral dissolvable powder - dosage 300mg no active ingredient
  Arms: Placebo

SUMMARY:
To determine the relief of GI discomfort after overfeeding with a high caloric meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without clinical diagnosed diseases with relevant effect on the gastrointestinal system or on visceral motility.
* Age ≥ 25 and ≤ 70 years
* BMI: 19-30 kg/m2
* Overall GI discomfort after high caloric meal of at least 5 on the VAS scale
* Male or female
* Written consent to participate in the study
* Subject is able and willing to follow the study protocol procedures
* If applicable, stable intake of chronic medication of at least 3 months

Exclusion Criteria:

Criteria for inclusion:

* Healthy volunteers without clinical diagnosed diseases with relevant effect on the gastrointestinal system or on visceral motility.
* Age ≥ 25 and ≤ 70 years
* BMI: 19-30 kg/m2
* Overall GI discomfort after high caloric meal of at least 5 on the VAS scale
* Male or female
* Written consent to participate in the study
* Subject is able and willing to follow the study protocol procedures
* If applicable, stable intake of chronic medication of at least 3 months

Criteria for exclusion:

* Relevant history, presence of any medical disorder (e.g. cancer, severe liver disease, severe renal disease, severe cardiovascular disease)
* Subject under prescription for medication for digestive symptoms such as anti-spasmodic, laxatives and anti-diarrheic drugs or use of PPI (proton pump inhibitors) or other digestive auxiliaries potentially interfering with this study at screening
* Intake of antibiotics in the last 4 weeks
* Women suffering from distinct PMS symptoms
* Acute gastrointestinal diseases including diarrhea and/or vomiting within the last 2 weeks
* Change of dietary habits within the 4 weeks prior to screening (for instance start of a diet high in fibers)
* Vegetarian or vegan nutrition style
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding subject.
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study.
* Participation in another clinical intervention study within the last 4 weeks and concurrent participation in another intervention clinical study
* Subject who according to the study staff's opinion is not suitable for participation in the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall gastrointestinal discomfort assessed with a visual analogue scale (VAS) | Chance over time after single dosage (pre, 0 minutes and after 5 minutes,15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes)
  In the current study, GI discomfort, following a high caloric meal, will be assessed with a visual analogue scale (VAS) before and after meal at defined timepoints.

SECONDARY OUTCOMES:
Assessment of gastrointestinal symptoms on a 6-point Likert scale | Chance over time after single dosage (pre, 0 minutes and after 5 minutes,15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes)
  In the current study, the following GI symptoms will be assessed: Feeling of fullness / tension, Passage of gas/ Flatulence, Bloating, GI discomfort, cramps, pain, Rumbling, Burping, Heartburn symptom, Nausea, Urge of defecate
Follow up assessment of gastrointestinal symptoms on a 6-point Likert scale | Day 1 immediately prior going to bed, day 2 immediately after wake up
  In the current study, the following GI symptoms will be assessed: Feeling of fullness / tension, Passage of gas/ Flatulence, Bloating, GI discomfort, cramps, pain, Rumbling, Burping, Heartburn symptom, Nausea, Urge of defecate, as well as overall gastrointestinal discomfort.
Monitoring of related adverse events | up to 14 hours after intake
  Reporting of adverse effects to evaluate tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Biotesys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No